CLINICAL TRIAL: NCT06959667
Title: Comparative Analysis of Nemonoxacin and Other Anti-methicillin Resistant Staphylococcus Aureus (Anti-MRSA) Antimicrobial Therapy in Patients With Complicated Skin and Soft Tissue Infections (cSSTI): a Retrospective Chart Review Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, WANG-HUEI SHENG, National Taiwan University Hospital
Other Study IDs: 202502099RIND
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Methicillin-susceptible S. Aureus (MSSA); Anti-methicillin Resistant Staphylococcus Aureus (Anti-MRSA); Complicated Skin and Soft Tissue,cSSTI
Keywords: methicillin-susceptible S. aureus (MSSA); Nemonoxacin; anti-methicillin resistant Staphylococcus aureus (anti-MRSA); complicated skin and soft tissue,cSSTI
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Use other antimicrobial therapy (vancomycin, teicoplanin, daptomycin, linezolid, or other anti-MRSA: Use other antimicrobial therapy (vancomycin, teicoplanin, daptomycin, linezolid, or other anti-MRSA antibiotics)
- Use Nemonoxacin: Use Nemonoxacin
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention
  Groups: Use Nemonoxacin

SUMMARY:
Increasing rates of antimicrobial resistant bacterial infections and antimicrobial therapy at home in elderly are great concern for medical care. The availability of new antibacterial agents that are effective against bacteria with resistance to other antibacterials is therefore critical to continued successful management of bacterial illnesses in the future. Nemonoxacin is a C-8 methoxy, non-fluorinated quinolone that retains potent broad-spectrum activities against Gram-positive and Gram-negative bacteria by selective inhibition of bacterial DNA topoisomerase.

Nemonoxacin had greater in-vitro activity against many Gram-positive bacteria, including methicillin-susceptible S. aureus (MSSA), and ciprofloxacin-susceptible and ciprofloxacin-resistant MRSA, levofloxacin-susceptible and levofloxacin-resistant S. pneumoniae, Streptococcus pyogenes, Streptococcus agalactiae, enterococci, and Enterobacterieacea species except Pseudomonas aeruginosa. Lowe selected mutation of Nemonoxacin, compared with other fluoroquinolones against antimicrobial resistant gram-positive bacteria had been reported.[5] Nemonoxacin could be used once-daily oral and intravenous formulations for the treatment of community-acquired pneumonia, including methicillin resistant Staphylococcus aureus (MRSA). However, nemonoxacin has less evidence of efficacy for complicated skin and soft tissue infection. In this retrospective study, we will investigate the treatment outcomes of nemonoxacin and compared with other anti-methicillin resistant Staphylococcus aureus (anti-MRSA) antimicrobial therapy in patients with complicated skin and soft tissue infections (cSSTI) by chart review.

ELIGIBILITY:
Inclusion Criteria:

* complicated skin and soft tissue (cSSTI) infection

Exclusion Criteria:

* no complicated skin and soft tissue (cSSTI) infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: complicated skin and soft tissue (cSSTI) infection
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical outcome of intravenous/oral nemonoxacin therapy compared with other antimicrobial therapy (vancomycin, teicoplanin, daptomycin, linezolid, or other anti-MRSA antibiotics) in patients with cSSTI. | between 01 January 2023 and 31 January 2025

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
To compare the clinical efficacy, antimicrobial efficacy, and adverse drug reactions of nemonoxacin in the treatment of complicated skin and soft tissue infections (cSSTIs) with other anti-MRSA antimicrobial therapies in patients with complicated skin and soft tissue infections.
Supporting Information: Study Protocol